CLINICAL TRIAL: NCT06705114
Title: Ultrasound Investigation of Tongue Movement During Mastication for Completely Edentulous Patients Rehabilitated by Mandibular Implant Retained Overdenture
Brief Title: Ultrasound Investigation of Tongue Movement for Implant Overdenture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A01010023RP
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-10

CONDITIONS: Prosthesis Durability
Keywords: Mastication; implant; mandibular; ultrasound; tongue movement
MeSH Terms: conditions — Prosthesis Failure | interventions — Denture, Complete

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group I: complete dentures (Active Comparator): Each patient received a newly constructed conventional complete denture.
  Interventions: Procedure: complete denture
- group II: mandibular implant overdenture (Active Comparator): Two dental implants were inserted in the patient's mandibular arch at the canine region using guided surgery and a delayed loading protocol.
  Interventions: Procedure: implant overdenture

INTERVENTIONS:
Procedure: complete denture — Each patient received a newly constructed conventional complete denture with optimal denture extension and lingualized balanced occlusal concept
  Arms: group I: complete dentures
Procedure: implant overdenture — Two dental implants were inserted in the patient's mandibular arch at the canine region using guided surgery and a delayed loading protocol.After 3-4 months, the dental implants were exposed and ball abutments were screwed into the implants. The housing of the ball attachments were incorporated into the fitting surface of the mandibular denture using a direct pick-up technique (Fig. 1B). The mandibular overdenture was then inserted into the patient's mouth and occlusal adjustment was done using articulating paper to remove any occlusal interferences. Follow-up visits were scheduled.
  Arms: group II: mandibular implant overdenture

SUMMARY:
This study aimed to examine the impact of mandibular implant overdentures on tongue movement during mastication.

DETAILED DESCRIPTION:
Each patient received a newly constructed conventional complete denture. To construct the radiographic stent, the mandibular denture was duplicated in clear acrylic resin and modified by placing multiple holes filled with radiopaque gutta-percha points. A stereolithographic surgical guide was then constructed using a dual scan technique with cone beam computerized tomography (CBCT, i-CAT Vision®, Imaging Sciences International, Hatfield, PA). Two dental implants were inserted in the patient's mandibular arch at the canine region using guided surgery and a delayed loading protocol. Patients were instructed to rinse their mouth with Chlorohexidine mouthwash just before the implant surgery and continue for one week. A prophylactic antibiotic (Amoxicillin and Clavulanic acid 125 mg) was administered one hour before the surgery and continued for one week after surgery. To control pain, a nonsteroidal anti-inflammatory drug (Ibuprofen 600 mg) was prescribed. After surgery, patients were prohibited from using the complete denture and were advised to follow a soft diet.

After one week, the mandibular denture was relieved and relined with soft relining material (Softliner; PROMEDICA) and delivered to the patient. After 3-4 months, the dental implants were exposed and ball abutments were screwed into the implants (Fig.1A). The housing of the ball attachments were incorporated into the fitting surface of the mandibular denture using a direct pick-up technique (Fig. 1B). The mandibular overdenture was then inserted into the patient's mouth and occlusal adjustment was done using articulating paper to remove any occlusal interferences. Follow-up visits were scheduled.

Tongue movement measurement The evaluation of tongue movement was conducted using an ultrasound imaging system (Toshiba Medical Systems Corporation, Tokyo, Japan) with a 3.1-MHz convex probe. A layer of ultrasound jelly (Sono Jelly, Toshiba Medical Systems Corporation) was applied to the patient's skin under the probe. The patient was instructed to sit in upright position, and the probe was placed under the chin area to allow the beam to pass through the distal surfaces of the second premolars on both the right and left sides. The probe was secured in place using a microphone stand (Panasonic System Networks Co., Ltd., Tokyo, Japan) with adjustable height and angle. The position of the tongue was confirmed on the B-mode image of the sagittal plane, which provided a two-dimensional recording of the slice through the oral cavity. The recording rate was 0.0476 seconds (21 frames per second). Ultrasound images were taken while the patient chewed 1/4 of a cookie in a normal manner until it was swallowed.

The ultrasound images were taken at two different oral conditions: 3 months after complete denture insertion and 3 months after mandibular implant overdenture insertion. The ultrasound data were exported from the imaging system via a USB port and transferred to a personal computer. The Articulate Assistant Advanced (AAA) software program version 221.2.0 was used to analyze the data. The software program provides a measurement fan, which is used to automatically set control points at the intersection of the tongue-surface spline and each radial axis. This is done using the AAA edge-detection algorithm, which detects dark-bright discontinuities in the image. (28) The spline was then fitted to the visible surface of the tongue in each relevant video frame (Fig. 2). From the start time (the beginning of mastication) to the end time (when the tongue moved up towards the palate at the start of swallowing), the tongue surface was traced in AAA.

The following items were measured:

1 -Duration of Chewing: From time of food ingestion to the time of beginning of first swallowing.

2- Cumulative displacement of the tongue during Chewing: The distance (in mm) from the tongue surface spline to the anchor point (A) was measured along the radial fan lines at three different points: 30 degrees posterior (B), the center (C), and 30 degrees anterior (D) (Fig. 3). This measurement process was repeated for consecutive video frames. The sum of absolute change between consecutive frames for all measurement points was detected.

3- Tongue surface shape during chewing.

ELIGIBILITY:
Inclusion Criteria:

* All patients were completely edentulous for at least one year, had a normal maxillo-mandibular relationship, and had available inter-arch space. They were nonsmokers and free from any systemic diseases that could affect implant osseointegration

Exclusion Criteria:

* Patients with head and neck surgery, skeletal deformity, and temporomandibular joint disorder were excluded from the study.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
ultrasound investigation of tongue movement | after 3 months of denture and overdenture insertion
  The evaluation of tongue movement was conducted using an ultrasound imaging system (Toshiba Medical Systems Corporation, Tokyo, Japan) with a 3.1-MHz convex probe. A layer of ultrasound jelly (Sono Jelly, Toshiba Medical Systems Corporation) was applied to the patient's skin under the probe. The patient was instructed to sit in upright position, and the probe was placed under the chin area to allow the beam to pass through the distal surfaces of the second premolars on both the right and left sides. The probe was secured in place using a microphone stand (Panasonic System Networks Co., Ltd., Tokyo, Japan) with adjustable height and angle. The position of the tongue was confirmed on the B-mode image of the sagittal plane, which provided a two-dimensional recording of the slice through the oral cavity. The recording rate was 0.0476 seconds (21 frames per second). Ultrasound images were taken while the patient chewed 1/4 of a cookie in a normal manner until it was swallowed.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry, mansoura university Mansoura, Egypt,, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Goncalves GSY, de Magalhaes KMF, Rocha EP, Dos Santos PH, Assuncao WG. Oral health-related quality of life and satisfaction in edentulous patients rehabilitated with implant-supported full dentures all-on-four concept: a systematic review. Clin Oral Investig. 2022 Jan;26(1):83-94. doi: 10.1007/s00784-021-04213-y. Epub 2021 Oct 13. PMID 34647147